CLINICAL TRIAL: NCT06669195
Title: Feasibility and Safety of Intravascular Lithotripsy for Acute Stent Under-expansion in Calcified Coronary Lesions
Brief Title: Intravascular Lithotripsy for Acute Stent Under-expansion in Calcified Coronary Lesions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuzhou Third People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-02-007-H01
Record Dates: First submitted 2024-10-31; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Coronary Artery Disease; Calcification
Keywords: Intravascular lithotripsy; stent under-expansion; calcified coronary lesions
MeSH Terms: conditions — Coronary Artery Disease; Calcinosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravascular lithotripsy group (Experimental)
  Interventions: Device: Intravascular lithotripsy group
- high-pressure balloon group (Active Comparator)
  Interventions: Device: high-pressure balloon group

INTERVENTIONS:
Device: Intravascular lithotripsy group — 20 subjects with stent under-expansion in calcified coronary lesions who met the inclusion/exclusion criteria were enrolled; subjects were assigned to the treatment group of Intravascular lithotripsy group.
  Arms: Intravascular lithotripsy group
Device: high-pressure balloon group — 20 subjects with stent under-expansion in calcified coronary lesions who met the inclusion/exclusion criteria were enrolled; subjects were assigned to the treatment group of high-pressure balloon group.
  Arms: high-pressure balloon group

SUMMARY:
Percutaneous coronary intervention (PCI) is the standard treatment for patients with coronary artery disease who have an indication for surgery. Coronary artery calcification not only makes stent delivery and expansion more difficult during PCI, but also increases the risk of vessel perforation. In addition, calcified plaque can lead to incomplete stent expansion, which increases the risk of in-stent restenosis and thrombosis. Although the technology and techniques of interventional devices continue to improve, heavily calcified lesions remain an important risk factor for PCI failure.

This study is a prospective, multicenter, randomized study. It is planned to select 40 cases of subjects with calcified plaque can lead to incomplete stent expansion who meet the inclusion/exclusion criteria. They are randomly dividing them into Intravascular lithotripsy treatment group and high-pressure balloon treatment group according to the ratio of 1:1. All subjects accept clinical follow-up after operation, at 30 days, 6 months, and 12 months after operation. Follow-up with angiography and OCT are conducted at 12 months. The primary endpoint was thickness of neointima at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Radiography inclusion criteria

  1. the angiography identified a severely calcified lesion with acute stent under-expansion, i.e., residual stenosis >20% after stenting and 16-atm dilatation with a post-dilatation balloon;
  2. target lesion stenosis must be ≥70% or ≥50% with clear evidence of myocardial ischaemia (visual assessment);
  3. target lesion vessel diameter is between 2.75mm and 4.0mm, target lesion length must be ≤30 mm (visual assessment);

General inclusion criteria

1. subjects at the age between ≥18 and ≤80 years old;
2. patients with symptoms or evidence of myocardial ischaemia;
3. subjects are willing to participate in the study, sign informed consent form, and accept clinical and angiography follow-up after PCI.

Exclusion Criteria:

* Radiography exclusion criteria

  1. in-stent lesions;
  2. For the left main disease and bifurcation lesion (branch vessel diameter shall be ≥ 2.5mm);
  3. Target lesions were total occlusive lesions (acute or chronic), long lesions (>30 mm), lesion vessel reference diameters >4.0 mm, and lesion angiomatous dilatation;

General inclusion criteria

1. Patients with severe congestive heart failure (NYHA Level IV severe heart failure) or severe valvular heart disease; or left ventricular ejection fraction of less than 35%;
2. Patients with stroke, peptic ulcer or gastrointestinal bleeding within the past 6 months; or patients with bleeding tendency or coagulation disorders;
3. Patients with severe liver failure (ALT and AST are larger than 3 times of the upper limit of normal value), who are judged to be not applicable to angiography by investigators;
4. Patients with severe renal failure(eGFR<30ml/minute) or such medical history, failure to comply with angiography conditions;
5. Subjects who are intolerance or allergic to heparin, contrast agent, Biolimus, polyethylene oxide and polylactic acid - glycolic acid polymer;
6. Patients who plans to accept selective operation within 1 year;
7. Patients who are participating in the clinical trial of other drug or device without reaching the time limit of primary endpoint;
8. Subjects who are considered to be not applicable to be enrolled by investigators due to other reasons.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-12 (Estimated); Primary Completion 2026-12-13 (Estimated); Study Completion 2027-03-13 (Estimated)

PRIMARY OUTCOMES:
the thickness of neointima | 12 months

IPD SHARING:
Plan to Share IPD: Undecided